CLINICAL TRIAL: NCT06484803
Title: Longitudinal Search for Neurobehavioral Underpins of Resilience to Stress
Brief Title: Resilience Among Trauma Survivors
Status: Enrolling by invitation | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: 0918-20-TLV
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: PTSD
Keywords: Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A major gap remains in understanding the neurobehavioral mechanism of individuals' variability in the dynamic process of responding to traumatic events. To address this gap, the proposed study is focused on two dominant survival processes: acute stress response and motivational behavior. Investigating the involvement of these processes in long-term recovery from a documented traumatic event, our study extends a prior longitudinal investigation in our lab that systematically assessed the neurobehavioral factors contributing to the development of PTSD.

DETAILED DESCRIPTION:
Individual responses to potentially traumatic stress exhibit wide variation, reflecting differences in stress resilience - denoting the capacity to adaptively cope with and recover from adversity (i.e. health despite adversity). To date, growing evidence tracing symptoms' changes following a potentially traumatic event has revealed distinct clinical trajectories, demonstrating variability in the individuals' recovery dynamics following a traumatic event. While some individuals regain homeostasis and recover over time, others experience chronic debilitating dysfunctions and exhibit long-term psychopathology. The current study aims to extend an original longitudinal investigation assessing recent trauma survivors three times within 14 months, with additional clinical and neurobehavioral assessment time points at ~80 months following the exposure to a documented traumatic event. While the previous study focused on assessing neurobehavioral indications of threat and reward sensitivity, this study specifically focused on acute stress response and motivational behavior with respect to trauma recovery trajectory.

Acute stress response involves immediate neurophysiological and psychological reactions to perturbing occurrence, transitioning from a reactive phase to a recovery phase. The reactivity phase is characterized by a threat to physical and mental homeostasis, manifested in multiple neurobiological processes. Subsequently, the stress response transitions to the recovery phase, distinguished by restoring homeostasis and establishing a new memory for coping in the future. The novel dataset collected in this study including fMRI task and resting state, behavioral and biological measurements, enables examination of the neurophysiological mechanism underlying lab-induced acute stress reactivity and recovery and associates it with long-term clinical outcomes following life event adversity. Motivation plays a crucial role in driving the individual's behavior toward a desirable (i.e. rewarding) goal and assists in adaptive coping with the environment. An intriguing finding in the original longitudinal study pointed to the importance of preserved reward processing for resilience. However, the study lacks an exploration of goal-based behavior in motivation which is critical for adaptive coping following stress (e.g. deciding to make an effort and pursue rewarding stimuli despite the possibility of encountering an unpleasant occurrence such as a traumatic reminder). In this project, we posit neurobehavioral aspects of motivational goal-directed behavior (as indicated by approaching or avoiding rewards under risk) will be associated with the long-term dynamics of recovery among trauma survivors. Neuronally, the indicated stress and motivation processes are depicted by functionality patterns in circuits involved in stress and threat (e.g. amygdala, insula, and periaqueductal gray; PAG), motivation (e.g. ventral striatum, orbital-PFC, and Ventral Tegmental Area; VTA) and memory, learning and emotion regulation (e.g. hippocampus and ventromedial-PFC).

In the current study, participants from the initial longitudinal study were recruited for a fourth-time point (~60 months following trauma exposure) and a fifth-time point (~80 months following trauma exposure). The fourth evaluation point involved clinical assessment, fMRI scan, physiological measurements, saliva collection for cortisol, and blood sampling (for epigenetic indices). The fifth time point involved home-based self-report questionnaires to evaluate the impact of the October 7th, 2023 events on the participants' clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the initial study after an exposure to a traumatic event.
* Age:18 - 70 years.
* Able to read and comprehend Hebrew.

Exclusion Criteria:

* Individuals who can't perform an MRI due to safety reasons (e.g. irremovable metals in their body) or claustrophobia.
* Individuals with a diagnosis of substance abuse, psychotic or bipolar I disorder.
* Individuals with documented head trauma with coma exceeding 30 minutes or with known neurological deficit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult civilians admitted to Tel-Aviv Sourasky Medical Center's Emergency Room (ER), following a potentially traumatic incident.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Clinical trajectories | Approximately 6 years
  Change in PTSD symptoms measured by change in Clinician-Administered PTSD Scale. The Clinician-Administered PTSD Scale is used to assess PTSD diagnostic status and symptom severity. We use both CAPS-V (according to DSM-4) and CAPS-5 (according to DSM-5) at 4 time points after exposure (1mo, 6mo, 14mo, ~60mo).
Change in PTSD symptoms following the October 7th, 2023 events | Half an hour
  Measured by the PTSD Checklist (PCL-5), a self-report measure (20 items) assessing the severity of PTSD symptoms, reflecting the diagnostic criteria of DSM-5. The PCL-5 total score can range from 0-80; with higher scores reflecting greater severity.
Change in anxiety symptoms following the October 7th, 2023 events | Half an hour
  Measured by the Beck Anxiety Inventory (BAI), a self-reported measure (21 items) of concurrent anxiety symptoms.
Change in depressive symptoms following the October 7th, 2023 events | Half an hour
  Measured by the Beck Depression Inventory (BDI), a self-reported measure (21 items) of depression symptoms and intensity, which was proven to be a good predictor of chronic PTSD at one week and one month after trauma.

SECONDARY OUTCOMES:
Neural response to acute stress induction and PTSD resilience | 4 hours
  During functional Magnetic Resonance Imaging (fMRI) session, an acute stress induction task known as The Montreal Imaging Stress Task (MIST) is administered. MIST is a psychosocial acute stress induction task incorporating mental arithmetic and social evaluation, tailored to the requirements of the fMRI environment. The task comprises three conditions: rest, training (control), and test (stress).
  The outcome will be measured as the changes in the salience network (e.g. amygdala, insula, ACC), default mode network (PCC, hippocampus), and central executive network (e.g. dorsolateral PFC), during acute stress induction vs control condition. These alterations will be correlated with Post-Traumatic Stress Disorder (PTSD) resilience, operationalized by the CAPS score.
Neural measures of reward and punishment and PTSD resilience | 4 hours
  A motivational task (Punishment, Reward, and Incentive Motivation Game; Primo) is conducted during an fMRI session. PRIMO is a dynamic motivational task designed to manipulate motivational aspects within the constraints of the fMRI environment. Neural measures of reward and punishment will be assessed during fMRI scanning. The region of interest (ROI) analysis of the ventral striatum (VS) and ventromedial prefrontal cortex (vmPFC) will be defined. Additionally, other mesolimbic nodes will be delineated based on a meta-analysis of reward-related literature. The outcome will be measured as the association between PTSD resilience, operationalized by the delta between the CAPS scores, and the contrast between reward vs punishment during the PRIMO task.
Neurobehavioral Measures of Approach-Avoidance Conflict Related to PTSD Resilience | 4 hours
  During the fMRI scanning session, neurobehavioral measures of approach-avoidance conflict will be evaluated as participants engage in the PRIMO task (see above). ROI analysis of the VS and ventral tegmental area (VTA) will be defined. Moreover, other mesolimbic nods will be defined based on a meta-analysis of approach-avoidance conflict. The outcome will be measured as the association between PTSD resilience, operationalized by the delta between the CAPS scores, and approach regions under high vs low goal conflict in the game (PRIMO).

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel